CLINICAL TRIAL: NCT02134652
Title: Ability of Bedside Ultrasound to Predict Progression of Severity of Disease in Dengue Fever
Status: Withdrawn | Type: Observational
Why Stopped: Unable to conduct study because of political issues in host country.
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Other Study IDs: EUS-3325
Record Dates: First submitted 2014-04-29; First posted 2014-05-09 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Dengue; Disease Progression
Keywords: Ultrasonography; World Health
MeSH Terms: conditions — Dengue; Disease Progression

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Suspected Dengue: Children with an acute febrile illness, and two of the following: headache, retro-orbital pain, myalgias, arthralgia, rash, hemorrhagic manifestations, or plasma leakage (i.e. shortness of breath, abdominal distention/pain) will all receive a diagnostic bedside ultrasound.
  Interventions: Other: diagnostic bedside ultrasound

INTERVENTIONS:
Other: diagnostic bedside ultrasound — Patients enrolled in this study will undergo bedside ultrasound during their initial presentation to the emergency department. Ultrasound imaging protocols include the following:
  * FAST Exam - Standard images will be obtained using the abdominal transducer. Images include the following: 1) sub-xyphoid 2)right upper quadrant (with right thorax) 3)left upper quadrant (with left thorax) and 4) suprapubic
  * Right Upper Quadrant Exam - Standard images will be obtained using the abdominal transducer. Images include the following: 1) Long axis of the gallbladder 2) Transverse axis of the gallbladder fundus 3) Transverse axis of the gallbladder body and 4) Transverse axis of the gallbladder neck.

SUMMARY:
The purpose of this study is determine the ability of bedide ultrasound performed in the Emergency Department and Outpatient Department can predict the severity of disease during a Dengue Fever outbreak in children, in Siem Reap, Cambodia. Our hypothesis is that the presence of gallbladder wall thickening and/or pleural effusions in children correlates with progression to Dengue hemorrhagic fever and Dengue shock. In addition, we hypothesize that sonographic imaging of pediatric patients presenting to the emergency department with a fever during a Dengue fever outbreak will change management and disposition.

DETAILED DESCRIPTION:
Dengue fever has various levels of severity, from mild disease to severe hemorrhagic complications and shock. Dengue is endemic world-wide and has been found in the United States. The mortality from dengue fever can be as high as 15-20%, with nearly 22,000 deaths annually, most of them children (Reddy, 2013). There is no reliable way to immediately predict which children presenting with a fever during a Dengue fever outbreak will progress to more severe disease. Some children with dengue fever will improve with limited clinical interventions, but others require intensive therapy. Limited healthcare resources in developing countries make decisions on treatment or disposition difficult as many children and poor clinical decision increase morbidity and mortality. In more developed countries such as the United States, early identification of patients with dengue fever has the potential to identify children who may benefit from early interventions. Identifying those patients is the first step in exploring early therapies to effect mortality. Previous research has demonstrated that intrathoracic/ peritoneal fluid and gallbladder wall thickening is associated with worsening of the clinical prognosis for hospitalized patients with dengue fever (Michels, 2013). We will explore earlier presentations in the emergency department and outpatient department.

Our hypothesis is that the presence of gallbladder wall thickening and/or pleural effusions in children correlates with progression to Dengue hemorrhagic fever and Dengue shock. In addition, we hypothesize that sonographic imaging of pediatric patients presenting to the emergency department with a fever during a Dengue fever outbreak will change management and disposition. Our specific aim is to 1) compare the accuracy of bedside ultrasound detection of intra-thoracic fluid, peritoneal free fluid, and gallbladder wall thickening and physical exam versus physical exam alone in diagnosing dengue fever and 2) determine the association between sonographic features of dengue (intra-thoracic fluid and gallbladder wall thickening) and clinical outcome in children with dengue fever.

This study is a prospective observational clinical study in the emergency department, inpatient ward, intensive care unit, and outpatient department of the Angkor Hospital for Children in Siem Reap, Cambodia. Study subjects will include children 16 years or less, who present during the annual Dengue Fever outbreak with suspected Dengue fever. Subjects include children with an acute febrile illness, and two of the following: headache, retro-orbital pain, myalgias, arthralgia, rash, hemorrhagic manifestations, or plasma leakage (i.e. shortness of breath, abdominal distention/pain). Clinicians will determine their clinical suspicion of dengue, intended therapeutic interventions and disposition following a history and physical exam but before ultrasound imaging. Study personnel will perform diagnostic bedside ultrasound imaging of the gallbladder and peritoneal and pleural spaces (FAST exam) and the clinician again determine their clinical suspicion of Dengue, intended therapeutic interventions and disposition. Patients will be followed to determine clinical outcome, therapeutic interventions and disposition. The primary endpoint is progression of disease. The secondary endpoint will be change in clinical care provided in the emergency department related to ultrasound imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Age >3 months and <16 years
2. Clinical suspicion of dengue hemorrhagic fever. (Revised WHO Classification System)
3. Not a prisoner or ward of the state
4. Parents able and willing to give consent. Children older then 7 able and willing to give assent

Exclusion Criteria:

1. Allergic to Ultrasound gel
2. Prisoners or wards of the state
3. Unstable patients
4. Known pleural effusion, ascites, or gallbladder wall thickening.

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study subjects will include children 16 years or less, who present during the annual Dengue Fever outbreak with suspected Dengue fever. Subjects include children with an acute febrile illness, and two of the following: headache, retro-orbital pain, myalgias, arthralgia, rash, hemorrhagic manifestations, or plasma leakage (i.e. shortness of breath, abdominal distention/pain)
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Progression of Disease | Patients who are discharged from home will be contacted a maximum of 10 days after discharge to acquire follow up data. Those patients who are admitted to the hospital will monitored for the entirety of their hospital stay, an average of about 2 weeks.
  Changes in clinical course or progression of disease in patients with Dengue Fever or Dengue Hemorrhagic Fever

SECONDARY OUTCOMES:
Clinical Care | Patients will receive an ultrasound in the emergency department or outpatient department. Within 2 hours of study enrollment, the treating physician will be made aware of the test results and will be queried for changes in decision making.
  Change in clinical care provided in the emergency department related to ultrasound imaging for patients presenting to the emergency department with symptoms of Dengue Fever.

OTHER OUTCOMES:
Disposition | Patients will receive an ultrasound in the emergency department or outpatient department. Within 2 hours of study enrollment, the treating physician will be made aware of the test results and will be queried for decision to admit versus discharge.
  Change in disposition related to ultrasound imaging in patients presenting to the emergency department with symptoms of Dengue Fever

CONTACTS AND LOCATIONS:
Overall Officials: Samuel D Licciardo, M.D., Principal Investigator — University of Massachusetts, Worcester; Romolo Gaspari, M.D., Ph.D., Study Chair — University of Massachusetts, Worcester
Locations (1):
- Angkor Hospital for Children, Siem Reap, Cambodia